CLINICAL TRIAL: NCT05804786
Title: Korean Multicenter Prospective Cohort of Diagnostic Bronchoscopy for Peripheral Lung Lesions
Brief Title: Prospective Cohort of Diagnostic Bronchoscopy for Peripheral Lung Lesions
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yeon Wook Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: K-ORIENT
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: Electromagnetic Navigation Bronchoscopy; Guided Bronchoscopy; Diagnosis; Radial Endobronchial Ultrasound
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group: Patients with peripheral pulmonary lesions which require histological differentiation because of the possibility of malignancy, and a biopsy can be attempted through guided bronchoscopy
  Interventions: Device: Guided bronchoscopy

INTERVENTIONS:
Device: Guided bronchoscopy — It is performed when a pulmonary lesion with a possibility of malignancy is found on chest CT and histological diagnosis and differentiation are required.
  Other Names: Device: Spin Thoracic Navigation System; Device: Radial EBUS probe

SUMMARY:
The primary objective is To evaluate the usefulness and safety of advanced guided bronchoscopy for histological diagnosis of peripheral pulmonary lesions.

The Secondary objective is to establish a strategy that can most effectively use endoscopes for early diagnosis of lung cancer in a real-world care environment by identifying patient/clinical/image/procedure-related characteristics that can optimize the practicality of emerging technologies.

DETAILED DESCRIPTION:
* Patients with peripheral pulmonary lesions who need histological diagnosis due to suspected lung cancer and whose lesions are judged capable of histological examination through guided bronchoscopy will be prospectively recruited.
* This study is a pure non-interventional pragmatic design. In addition to biopsy for lung lesions using bronchoscopy, lung cancer staging and tests necessary for metastases and treatment for diagnosed lung cancer are performed according to existing guidelines and the judgment of medical staff.
* We will analyze the clinical characteristics of guided bronchoscopy procedures used in clinical practice and the main results during the follow-up period of up to one year (diagnostic yield, sensitivity, safety, practicality, and various factors affecting usefulness).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agreed in writing to participate in this study
2. Adult men and women over 19 years of age
3. Patients who visited the hospital with lung lesions suspected of lung cancer and require a diagnostic biopsy
4. Patients capable of biopsy through guided bronchoscopy

Exclusion Criteria:

1) Patients who are unable to express their opinions and cannot cooperate due to a lack of cognitive function

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral pulmonary lesions that require histological differentiation because of the possibility of malignancy and are scheduled for biopsy attempted through guided bronchoscopy
Sampling Method: Probability Sample
Enrollment: 1240 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield at index | Upon reports of pathologic results (up to 2 weeks after bronchoscopy)
  The proportion of pathologic results that leads to a specific malignant or benign

SECONDARY OUTCOMES:
Diagnostic accuracy at 12 months | Confirmed by follow-up results at 1 year
  True positive + True negative (confirmed benign with follow-up of at least 1yr without progression) / Total procedures
  Pathologic results of a malignant or benign specific diagnosis based on the samples collected via index ENB procedure are categorized as true positives or true negatives.
  For pathologic results of a benign non-specific diagnosis and non-diagnostic results, follow-up data would be used to determine whether the 12-month status corroborates the benign results. Based on definition scenarios, these results will be determined as true negatives or false negatives. Diagnostic yields based on different scenarios will be reported.
Sensitivity for malignancy | Confirmed by follow-up results at 1 year
  True positive/Confirmed malignancy cases
Complication | Confirmed by follow-up results at 1 year
  Evaluate complications due to guided bronchoscopic biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Wook Kim, MD., PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (11):
- South Korea (11):
  - Dongsan Hospital Keimyung University School of Medicine, Daegu
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Chunnam National University Hwasun Hospital, Hwasun
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Gangnam Severence Hospital, Seoul
  - Hanyang University Hostpital, Seoul
  - The Catholic University of Korea, Seoul, Korea, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folch EE, Pritchett MA, Nead MA, Bowling MR, Murgu SD, Krimsky WS, Murillo BA, LeMense GP, Minnich DJ, Bansal S, Ellis BQ, Mahajan AK, Gildea TR, Bechara RI, Sztejman E, Flandes J, Rickman OB, Benzaquen S, Hogarth DK, Linden PA, Wahidi MM, Mattingley JS, Hood KL, Lin H, Wolvers JJ, Khandhar SJ; NAVIGATE Study Investigators. Electromagnetic Navigation Bronchoscopy for Peripheral Pulmonary Lesions: One-Year Results of the Prospective, Multicenter NAVIGATE Study. J Thorac Oncol. 2019 Mar;14(3):445-458. doi: 10.1016/j.jtho.2018.11.013. Epub 2018 Nov 23. PMID 30476574
- [Background] Ost DE, Ernst A, Lei X, Kovitz KL, Benzaquen S, Diaz-Mendoza J, Greenhill S, Toth J, Feller-Kopman D, Puchalski J, Baram D, Karunakara R, Jimenez CA, Filner JJ, Morice RC, Eapen GA, Michaud GC, Estrada-Y-Martin RM, Rafeq S, Grosu HB, Ray C, Gilbert CR, Yarmus LB, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic Yield and Complications of Bronchoscopy for Peripheral Lung Lesions. Results of the AQuIRE Registry. Am J Respir Crit Care Med. 2016 Jan 1;193(1):68-77. doi: 10.1164/rccm.201507-1332OC. PMID 26367186
- [Background] Folch EE, Labarca G, Ospina-Delgado D, Kheir F, Majid A, Khandhar SJ, Mehta HJ, Jantz MA, Fernandez-Bussy S. Sensitivity and Safety of Electromagnetic Navigation Bronchoscopy for Lung Cancer Diagnosis: Systematic Review and Meta-analysis. Chest. 2020 Oct;158(4):1753-1769. doi: 10.1016/j.chest.2020.05.534. Epub 2020 May 23. PMID 32450240
- [Background] Vachani A, Maldonado F, Laxmanan B, Kalsekar I, Murgu S. The Impact of Alternative Approaches to Diagnostic Yield Calculation in Studies of Bronchoscopy. Chest. 2022 May;161(5):1426-1428. doi: 10.1016/j.chest.2021.08.074. Epub 2021 Sep 7. No abstract available. PMID 34506792
- [Background] Bowling MR, Kohan MW, Walker P, Efird J, Ben Or S. The effect of general anesthesia versus intravenous sedation on diagnostic yield and success in electromagnetic navigation bronchoscopy. J Bronchology Interv Pulmonol. 2015 Jan;22(1):5-13. doi: 10.1097/LBR.0000000000000120. PMID 25590477
- [Background] Kops SEP, Heus P, Korevaar DA, Damen JAA, Idema DL, Verhoeven RLJ, Annema JT, Hooft L, van der Heijden EHFM. Diagnostic yield and safety of navigation bronchoscopy: A systematic review and meta-analysis. Lung Cancer. 2023 Jun;180:107196. doi: 10.1016/j.lungcan.2023.107196. Epub 2023 Apr 19. PMID 37130440